CLINICAL TRIAL: NCT00150215
Title: An Oral, Rising Single-Dose Tolerance, Pharmacokinetic, and Pharmacodynamic Study of Pf-00184562 Capsules In Healthy Volunteers
Brief Title: A First In Human Study Of PF-00184562 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: PPD Development, LP (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A6241001
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2006-07-25 (Estimated); Status verified 2006-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

INTERVENTIONS:
Drug: PF-00184562
Drug: Olanzapine

SUMMARY:
The purposes of this study are:

* To determine the safety, tolerability and pharmacokinetics of single doses of PF-00184562; and
* To explore the exposure-response relationship of neuropsychometric and tolerability measures of PF-00184562 compared to olanzapine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects of non-childbearing potential

Exclusion Criteria:

* Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, pancreatic, psychiatric, neurologic, active infections, immunological, or allergic disease (including drug allergies and seasonal allergies at time of dosing).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18
Dates: Start 2005-07; Study Completion 2005-10

PRIMARY OUTCOMES:
Safety and tolerability of single dose PF-00184562 as determined by: adverse event reporting, clinical laboratory results, vital signs, physical examinations, and electrocardiograms (ECGs).
Pharmacokinetic profile of PF-00184562 maximum concentration (Cmax)
Time to obtain maximum concentration (tmax), area under concentration-time curve (AUC), and terminal half-life (t1/2).
Exposure-response relationship of neuropsychometric and tolerability measures of PF-00184562 compared to olanzapine.
All measurements to be assessed over single doses.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Austin, Texas, United States